CLINICAL TRIAL: NCT00348400
Title: Brimonidine Purite 0.15% Versus Dorzolamide 2% Used as Adjunctive Therapy to Latanoprost
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 5099
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2007-06-01 (Estimated); Status verified 2007-05

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Brimonidine Tartrate; dorzolamide; Latanoprost

INTERVENTIONS:
Drug: Brimonidine Purite 0.15%, Dorzolamide 2%, Latanoprost

SUMMARY:
Evaluate the relative efficacy and tolerability of Alphagan P compared to Trusopt as adjunctive therapy

ELIGIBILITY:
Inclusion Criteria:

* · Male or female > 18 years of age

  * Diagnosis of open-angle glaucoma or ocular hypertension
  * IOP > 16 mm Hg in each eye at the latanoprost -treated baseline evaluation
  * Presently on latanoprost monotherapy for at least 6 weeks
  * Ability to provide informed consent and likely to complete all study visits

Exclusion Criteria:

* · Known contraindication or allergy to brimonidine or any of its components

  * Subjects must be naive to brimonidine 0.2% or brimonidine Purite 0.15% and dorzolamide 2%
  * Uncontrolled systemic disease
  * Active ocular disease other than glaucoma or ocular hypertension (e.g. uveitis, ocular infections, or severe dry eye). Patients with chronic mild blepharitis, cataract, age-related macular degeneration, or background diabetic retinopathy may be enrolled at the discretion of the investigator.
  * Required use of ocular medications other than the study medications during the study (intermittent use of artificial tear product is allowed).
  * Corneal abnormalities
  * History of intraocular surgery within the last 3 months
  * Female patients of childbearing potential who are pregnant, lactating, planning a pregnancy, or not using a reliable form of birth control
  * Visual field loss, which in the opinion of the investigator, is functionally significant, or evidence of progressive visual field loss within the last year.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Robert Noecker, MD, Principal Investigator — UPMC Eye Center
Locations (1):
- Dr. Noecker, Pittsburgh, Pennsylvania, United States